CLINICAL TRIAL: NCT06802978
Title: Study of Lipid Profile in Diabetic and Non Diabetic Chronic Kidney Disease Patients in Sohag University Hospital
Brief Title: Lipid Profile in Diabetic and Non Diabetic CKD Patients
Acronym: CKD
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shaimaa Mahmoud Elsayed Abdel-Raheem, Principal investigator resident at the Internal Medicine Department, Sohag University Hospital, Sohag University
Other Study IDs: Soh-Med--25-1-07MS
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic CKD patients: This group includes participants aged over 20 years who have been diagnosed with both chronic kidney disease (CKD) and diabetes mellitus.
- Non-diabetic CKD patients: participants aged over 20 years who have been diagnosed with chronic kidney disease (CKD) but do not have a current or past diagnosis of diabetes mellitus.

SUMMARY:
The goal of this observational study is to compare blood lipid (fat) levels in participants with chronic kidney disease (CKD) with diabetes and without diabetes and who over 20 years old.

The main question this study aims to answer is:

Does having diabetes make fat problems worse in people with chronic kidney disease (CKD), or is there no connection between them?

Researchers will compare the blood lipid (fat) levels in people with chronic kidney disease (CKD) who have diabetes and those without diabetes to see if having diabetes makes lipid problems worse in CKD patients, or if there is no connection between diabetes and changes in lipid levels.

Participants will need to fast for 10 hours before undergoing this test. This means not eating any food or drinking anything except water.

Samples will be taken and sent to laboratory immediately.

ELIGIBILITY:
Inclusion Criteria:

* Patients of chronic kidney disease (CKD) presenting to the Sohag University Hospital
* Patients aged above 20 years of age.
* All patients who have given consent for enrolling into the study.

Exclusion Criteria:

* Patients aged 20 years of age or below.
* Patients on lipid-lowering drugs.
* Kidney transplanted patients.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met all the inclusion criteria were selected randomly. No distinction is made between males and females.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Assessment and comparison of the lipid profile between diabetic and non-diabetic chronic kidney disease patients using the colorimetric method on a fully automated biochemistry analyser. | February 2025 to May 2025.
  Lipid profile were assessed in samples of chronic kidney disease patients , both with diabetes and without diabetes, after obtaining informed consent to compare lipid profile between these two groups.
  Overnight fasting samples were taken and sent to the laboratory immediately. Serum was separated within 2 hours after collection to prevent artifactual changes in the concentration of HDL. After clot retraction occurred, the serum was transferred to a centrifuge tube and centrifuged at 2000 rpm for 5 minutes. The clear supernatant serum was then pipetted out using dry piston pipettes with disposable tips and stored in dry thin walled vials at 4°C. The samples were analyzed on the same day.
  The following parameters were analyzed using the colorimetric method on a fully automated biochemistry analyser.
  1. Serum Cholesterol
  2. Serum Triglyceride
  3. Serum HDL (high-density lipoprotein)
  4. Serum LDL ( low-density lipoprotein)
  5. Serum VLDL (very low-density lipoprotein)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine , Sohag University Hospital., Sohag, Egypt